CLINICAL TRIAL: NCT04862988
Title: Reliability and Validity of Urdu Version of Global Physical Activity Questionnaire (GPAQ-U)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00233
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Physical Activity
Keywords: GPAQ; reliability,; Validity; Urdu
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The GPAQ questionnaire is used to measure the physical activity. In this study, Investigators will observe the reliability and validity of global physical activity questionnaire in Urdu language in Pakistan among students to assess physical activity.

DETAILED DESCRIPTION:
The aim of study is to translate and culturally adapt Global physical Activity Questionnaire (GPAQ) into Urdu language and secondly to investigate the reliability and validity of GPAQ in Pakistan among university students. This study will be cross sectional survey study in which convenience sampling technique will be used.

The results of study will help to know the validity and reliability of GPAQ in Urdu version among students in Pakistan. The reliability of the questionnaire will be checked through internal consistency and test-retest methods. Internal consistency will be analyzed with Cronbach's alpha value. Test-retest reliability will be assessed using an intra-class correlation coefficient with 100 patients

ELIGIBILITY:
Inclusion Criteria:

- Male and female aged over 18 years Pakistani national and native Urdu speakers Able to read and understand Urdu Studying in University level

Exclusion Criteria:

Male or female having any disability Any recent illness or any injury

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students, because they are usually engaged in their studies and have no enough time to do any physical activity resulting in decline in their overall health status.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Global Physical Activity Questionnaire (GPAQ) | 1st day
  A measuring instrument to evaluate the duration of vigorous and moderate physical activities that are performed in daily living routine. Each object has a specific code starting from P1 to P16 and then activity is calculated in MET value. For Work and Recreational domains, Moderate MET value is 4.0 and Vigorous MET value is 8.0 while for Transport domains MET value is 4.0
Global Physical Activity Questionnaire (GPAQ) | 2nd day
  A measuring instrument to evaluate the duration of vigorous and moderate physical activities that are performed in daily living routine. Each object has a specific code starting from P1 to P16 and then activity is calculated in MET value. For Work and Recreational domains, Moderate MET value is 4.0 and Vigorous MET value is 8.0 while for Transport domains MET value is 4.0

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 1st day
  A questionnaire for the assessment of population surveillance of physical activity among the adults having age(15-69).
  Expressed as MET-minutes per week: MET level x minutes of activity/day x days per week

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No